CLINICAL TRIAL: NCT05686655
Title: Sleep Quality Among Children And Adolescents With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amal Mohamed Abdelwahab, resident at pediatric departement at el helal hospital, Sohag University
Other Study IDs: soh-Med-22-12-05
Record Dates: First submitted 2023-01-09; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetes children
  Interventions: Other: questionnaire about sleep quality in diabetic children

INTERVENTIONS:
Other: questionnaire about sleep quality in diabetic children — Pittsburgh sleep quality index

SUMMARY:
Sleep is an important health behavior for children and adolescents due to the impact it has on both mental and physical development. Although sleep is considered a resting period, it is also a period when the brain work to encode and consolidate memories into more stable representations for long term recall . Unfortunately, pediatric sleep disorders affect 25 - 40% of youth and several studies showed that children with chronic illness experience more problems with initiating and maintaining sleep than their non- chronically ill children .

Type 1 diabetes mellitus (T1DM) affects the quality of sleep in children and adolescents as well as their caregivers. Sleep disturbances in patients with T1DM may negatively impact their ability to manage their diabetes .

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 6 to 15 years .
* diagnosed with T1DM for at least 6 months
* attending the pediatric diabetes outpatient clinic at Sohag University Hospital.
* Age and sex matched control group for acute non-serious illnesses

Exclusion Criteria:

* Children and adolescents with associated neurological or psychiatric disorders .

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Children and adolescents aged 6 to 15 years diagnosed with T1DM for at least 6 months and attending the pediatric diabetes outpatient clinic at Sohag University Hospital will be included in the study.
  Age and sex matched control group will be included from children and adolescents attending the general pediatric outpatient clinic at Sohag University hospital for acute non-serious illnesses.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
duration of nighttime sleep in hours in night times and weekends | in the past month
  duration of nighttime sleep in hours in night times and weekends
sleep problems as frequent awakening during the night | in the past month
  sleep problems as frequent awakening during the night

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reutrakul S, Thakkinstian A, Anothaisintawee T, Chontong S, Borel AL, Perfect MM, Janovsky CC, Kessler R, Schultes B, Harsch IA, van Dijk M, Bouhassira D, Matejko B, Lipton RB, Suwannalai P, Chirakalwasan N, Schober AK, Knutson KL. Sleep characteristics in type 1 diabetes and associations with glycemic control: systematic review and meta-analysis. Sleep Med. 2016 Jul;23:26-45. doi: 10.1016/j.sleep.2016.03.019. Epub 2016 Jun 8. PMID 27692274
- [Background] Monzon A, McDonough R, Meltzer LJ, Patton SR. Sleep and type 1 diabetes in children and adolescents: Proposed theoretical model and clinical implications. Pediatr Diabetes. 2019 Feb;20(1):78-85. doi: 10.1111/pedi.12797. Epub 2018 Dec 4. PMID 30447038
- [Background] Turner SL, Queen TL, Butner J, Wiebe D, Berg CA. Variations in Daily Sleep Quality and Type 1 Diabetes Management in Late Adolescents. J Pediatr Psychol. 2016 Jul;41(6):661-9. doi: 10.1093/jpepsy/jsw010. Epub 2016 Mar 19. PMID 26994852
- [Background] Suleiman KH, Yates BC, Berger AM, Pozehl B, Meza J. Translating the Pittsburgh Sleep Quality Index into Arabic. West J Nurs Res. 2010 Mar;32(2):250-68. doi: 10.1177/0193945909348230. Epub 2009 Nov 14. PMID 19915205